CLINICAL TRIAL: NCT05754749
Title: Comparison of Contrast Enhanced Digital Breast Tomosynthesis and Magnetic Resonance Imaging in Patients With Known Breast Lesions
Brief Title: Comparison of CE-DBT and MRI in Patients With Known Breast Lesions
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC2139
Record Dates: First submitted 2023-02-21; First posted 2023-03-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Iohexol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contrast-enhanced digital breast tomosynthesis (CE-DBT) (Experimental): Participants with known breast lesions will be imaged using contrast-enhanced digital breast tomosynthesis (CE-DBT) with Iohexol 350 mg I/mL.
  Interventions: Drug: Iohexol 350 Mg/mL Injectable Solution

INTERVENTIONS:
Drug: Iohexol 350 Mg/mL Injectable Solution — Participants will be scanned with the digital breast tomosynthesis (DBT) system before and after the intravenous administration of iodinated contrast agent, iohexol 350mg I/mL at a dose of 1.5 mL/kg body weight. Images will be acquired of the breast of interest prior to the administration of contrast, followed by at approximately 2 minutes and 5 minutes after administration. For the purposes of this study, imaging will focus on a single breast to simplify data acquisition.
  Other Names: Contrast- enhanced digital breast tomosynthesis (CE-DBT)

SUMMARY:
The purpose of this pilot study is to compare radiologist confidence level in evaluating patients with known breast lesions between contrast enhanced digital breast tomosynthesis (CE- DBT) and contrast enhanced dynamic magnetic resonance imaging (CE-MRI) acquired as a part of a standard clinical workup.

DETAILED DESCRIPTION:
This is a pilot study of CE-DBT scans to evaluate its utility relative to breast CE-MRI. Twenty women who have planned or received conventional breast MRI imaging at UNC Hospitals will be recruited for the study. Participants will be scanned with the DBT system after the administration of iodinated contrast agent. Images will be acquired prior to the administration of contrast, followed by at approximately 2 minutes and 5 minutes. For the purposes of this study, imaging will focus on a single breast to simplify data acquisition.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years old
* Planned or received conventional breast MRI at UNC Hospitals within 3 months prior to or after the research scan
* Suspected breast lesion based on prior imaging (BIRADS 4 or greater)
* Able to provide written informed consent

Exclusion Criteria:

* Severe untreatable claustrophobia
* Implanted metallic devices, parts, vascular clips, or other foreign bodies (including breast implants)
* Known hypersensitivity to iodinated contrast agent or to any component of iodinated contrast refractory to standard medications (antihistamines, steroids)
* Impaired kidney function (serum creatinine level > 1.8 mg/dl or a glomerular filtration rate < 60 as approximated using serum creatinine levels within the last 30 days prior to the research scan) unless anuric and on dialysis
* Any woman who is pregnant or has reason to believe she is pregnant (the possibility of pregnancy has to be excluded by negative urine β-HCG results, obtained within 24 hours prior to the research scan, or on the basis of patient history, as defined by the UNC IRB SOP 4801)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-08-22 (Estimated); Study Completion 2026-08-22 (Estimated)

PRIMARY OUTCOMES:
Reader confidence in identifying lesions on CE-DBT compared to contrast enhanced dynamic breast MRI (arbitrary units) | Calculated once all imaging is complete [Anticipated 1.5 years]
  To compare (using a reader study) the reader confidence in identifying lesions on CE-DBT to the reader confidence in identifying lesions on contrast enhanced dynamic breast MRI.

SECONDARY OUTCOMES:
Contrast enhancement curves of CE-DBT compared to conventional MRI (arbitrary units) | Calculated once all imaging is complete [Anticipated 1.5 years]
  To compare (using a reader study) the contrast enhancement curves of CE-DBT to the contrast enhancement curves of contrast enhanced dynamic breast MRI in evaluation of known breast lesions for predicting malignancy.
Diagnostic accuracy of CE-DBT compared to contrast enhanced dynamic breast MRI (arbitrary units) | Calculated once all imaging is complete [Anticipated 1.5 years]
  To compare (using a reader study) the diagnostic accuracy of CE-DBT to the diagnostic accuracy of contrast enhanced dynamic breast MRI in evaluation of known breast lesions for predicting malignancy.
Sensitivity of CE-DBT compared to contrast enhanced dynamic breast MRI (arbitrary units) | Calculated once all imaging is complete [Anticipated 1.5 years]
  To compare (using a reader study) the sensitivity of CE-DBT to the sensitivity of contrast enhanced dynamic breast MRI in evaluation of known breast lesions for predicting malignancy.
Specificity of CE-DBT compared to contrast enhanced dynamic breast MRI (arbitrary units) | Calculated once all imaging is complete [Anticipated 1.5 years]
  To compare (using a reader study) the specificity of CE-DBT to the specificity of contrast enhanced dynamic breast MRI in evaluation of known breast lesions for predicting malignancy.
Positivity predictive value of CE-DBT compared to contrast enhanced dynamic breast MRI (arbitrary units) | Calculated once all imaging is complete [Anticipated 1.5 years]
  To compare (using a reader study) the positivity predictive value of CE-DBT to the positivity predictive value of contrast enhanced dynamic breast MRI in evaluation of known breast lesions for predicting malignancy.
Receiver Operating Characteristic (ROC) curves of CE-DBT compared to contrast enhanced dynamic breast MRI (arbitrary units) | Calculated once all imaging is complete [Anticipated 1.5 years]
  To compare (using a reader study) the ROC curves of CE-DBT to the ROC curves of contrast enhanced dynamic breast MRI in evaluation of known breast lesions for predicting malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hitt, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.